CLINICAL TRIAL: NCT02462941
Title: Prospective Analysis of Low-Dose Adenosine on Sinus and Atrioventricular Nodal Conduction in the Pediatric Transplanted Heart
Brief Title: Analysis of Adenosine on Sinus and Atrioventricular Nodal Conduction in the Pediatric Transplanted Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Eric Silver, Assistant Professor of Pediatrics at the Columbia University Med, Dept of Pediatrics Cardiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAO8054
Record Dates: First submitted 2015-02-26; First posted 2015-06-04 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Sinus Bradycardia; Atrioventricular Block
Keywords: Heart transplant; Adenosine; Pediatrics
MeSH Terms: conditions — Atrioventricular Block | interventions — Adenosine; Cardiac Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adenosine (Experimental): After cardiac catheterization, the study protocol will begin with 12.5µg/kg of adenosine (one eighth the recommended starting clinical dose), and will double to 25µg/kg, 50µg/kg, 100µg/kg and finally 200µg/kg (not to surpass the total maximum dose of 12mg). A pacing catheter will be placed within the right ventricle prior to medication administration. Escalating doses will stop if ventricular pacing is required due to a ventricular pause greater than 12 seconds or if atrioventricular block is demonstrated with a ventricular pause less than 12 seconds. If there is no prolonged pause requiring pacing and no demonstration of medication effect the subsequent dose will be given.
  Interventions: Drug: Adenosine; Procedure: Cardiac catheterization

INTERVENTIONS:
Drug: Adenosine — Testing escalating doses of adenosine in pediatric heart transplant patients
  Other Names: No brand names
Procedure: Cardiac catheterization — (non-experimental) standard procedure

SUMMARY:
Heart transplants save the lives of nearly 500 children in heart failure per year. Columbia is one of the largest pediatric heart transplant centers in the world, averaging 25 transplants per year, and providing ongoing care to nearly 250 children with transplanted hearts. After transplant, children are at increased risk to develop sudden onset of abnormally fast heart rates. This research project will study adenosine, a medication that is routinely used to slow fast heart rates in non-transplanted children (i.e. normal hearts), and its effects on the transplanted heart. Adenosine is often not used in patients with transplanted hearts because, based on prior limited research in adult patients, the standard adult dose may have a longer medication effect, producing a slower heart rate for an undesirable period of time. However, the current alternatives to adenosine treatment are either inappropriate for the pediatric age range, or have increased risk of unwanted side effects. This research project will answer two questions: is adenosine safe to give a child who has had a heart transplant, and will it be effective in treating the fast heart rate?

All pediatric heart transplant patients undergo regular heart testing, known as a cardiac catheterization, one or more times per year. Three days before testing, participants will be asked to stop a regular medication, dipyridamole, because it slows the breakdown of adenosine in the body, and may increase its effects. (Of note, all patients that are on dipyridamole are also on aspirin, which gives a second line of heart protection, and will not be stopped.) After regular cardiac catheterization, all patients will already have intravenous (IV) access to give medication. Also, this setting allows the opportunity to have a back-up pacing catheter in the heart, ensuring that there will not be a longer than desired effect from the medication. Adenosine will be given per a low-dose protocol until either the medication effect is seen or the maximum dose is reached. There will be no difference in procedure recovery period time, and patients will resume regular home medications after finishing the test. As Columbia is one of largest pediatric heart transplant centers in the world, studying the effects of adenosine at low doses will benefit the investigators population greatly, either to find a new recommended medication dose, or to provide evidence that this medication is truly inadvisable for the investigators patients.

The initial study was completed with all 80 patients enrolled and tested. Subsequent testing is now ongoing on patients in whom dipyridamole was stopped prior to their initial testing with a repeat study without discontinuing the dipyridamole. We anticipate re-testing about 30 of the 80 patients.

DETAILED DESCRIPTION:
After cardiac catheterization, the study protocol will begin with 12.5µg/kg of adenosine (one eighth the recommended starting clinical dose), and will double to 25µg/kg, 50µg/kg, 100µg/kg and finally 200µg/kg (not to surpass the total maximum dose of 12mg). A pacing catheter will be placed within the right ventricle prior to medication administration. Escalating doses will stop if ventricular pacing is required due to a ventricular pause greater than 12 seconds or if atrioventricular block is demonstrated with a ventricular pause less than 12 seconds. If there is no prolonged pause requiring pacing and no demonstration of medication effect the subsequent dose will be given.

Progression to the next dose of the adenosine will depend on both the primary and secondary study outcomes. If the adenosine dose produces clinically significant bradycardia (> 12 seconds), ventricular pacing will be used to maintain cardiac output, and the dose will be considered unsafe to use clinically and testing will end for that patient. If the adenosine dose produces atrioventricular block but with a pause of less than 12 seconds (thus does not require pacing), the dose will be considered effective and the study will terminate as well. However, if the adenosine dose does not produce atrioventricular block or require pacing intervention, the dose will be considered safe but ineffective and the study will progress to the next higher dose. Before dose progression, the study will pause for additional 30 seconds to ensure complete adenosine metabolism, as the half-life of adenosine is less than 10 seconds and does not exhibit cumulative effects. The subsequent dose will then be administered and the ECG observed for clinically significant bradycardia and atrioventricular block. This will be repeated until clinically significant bradycardia and/or atrioventricular block is observed, or up to the final 200μg/kg (not to surpass the total maximum of 12mg) dose.

The same study protocol is being utilized to retest the subset of patients in whom dipyridamole was discontinued prior to the initial testing to further understand the safety of administering adenosine to heart transplant patients chronically maintained on dipyridamole.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a heart transplantation and who receive their routine care at the Morgan Stanley Children's Hospital of New York, Columbia University Medical Center

Exclusion Criteria:

* Patients admitted to the inpatient heart failure team
* Patients present for their first outpatient catheterization after new transplant
* Abnormal hemodynamics concerning for acute rejection
* Patients present for follow up of rejection (last biopsy positive)
* Ingested methylxanthine-containing foods that day
* Patients taking oral dipyridamole and did not discontinue it 3 days prior to testing
* Prior transplant history of coronary artery vasculopathy with this allograft or concern for abnormal coronary vasculature by angiography on the day of the catheterization
* Patients taking carbamazepine (may potentiate adenosine effect)
* Patients with known conduction disease (first, second or third degree atrioventricular block) and/or with pre-existing sinus node dysfunction (based on pre-existing ECG, Holter or inpatient telemetry)
* Patients/guardians unable to give consent in English

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Incidence of sinus bradycardia or atrioventricular block with low-dose adenosine administration that is greater than 12 seconds and requires hemodynamic intervention (ventricular escape pacing). | Up to 1 hour after the catheterization

SECONDARY OUTCOMES:
Prevalence of inducing atrioventricular block (defined as a single non-conducted P wave) at adenosine doses lower than suggested starting dose (100µg/kg) in PALS algorithm. | Up to 1 hour after the catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Silver, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Flyer JN, Zuckerman WA, Richmond ME, Anderson BR, Mendelsberg TG, McAllister JM, Liberman L, Addonizio LJ, Silver ES. Prospective Study of Adenosine on Atrioventricular Nodal Conduction in Pediatric and Young Adult Patients After Heart Transplantation. Circulation. 2017 Jun 20;135(25):2485-2493. doi: 10.1161/CIRCULATIONAHA.117.028087. Epub 2017 Apr 27. PMID 28450351